CLINICAL TRIAL: NCT04437628
Title: Prognostic Value Of Short-Term Follow-up Biomarkers After Discharge In hOspitalized Patients With Acute Heart Failure
Acronym: POSTBIO-HF
Status: Recruiting | Type: Observational
Sponsor: Wonju Severance Christian Hospital (Other)
Collaborators: Roche diagnostics Korea (Unknown)
Responsible Party: Principal Investigator, Byung-Su Yoo, Professor, Wonju Severance Christian Hospital
Other Study IDs: CR320021
Record Dates: First submitted 2020-06-16; First posted 2020-06-18 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Heart Failure
Keywords: Heart failure; Biomarkers; Prognosis
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Biospecimen Retention: None Retained — Blood sample for biomarker analysis (NP and GDF-15) within 30 days and at 6 months (±1 month) after discharge
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Several surrogate biomarkers including natriuretic peptide(NP), and growth differentiation factor-15(GDF-15) and ST2 has prognostic significance in heart failure(HF), and reductions in its value may predict clinical improvement. However, there are limited data regarding the prognostic value of these biomarkers during short-term follow-up after discharge in acute decompensated heart failure. The purpose of this study is to evaluate the prognostic value of short-term follow-up surrogate biomarkers for predicting prognosis of hospitalized patients with acute decompensated heart failure.

ELIGIBILITY:
Inclusion Criteria: the diagnosis of Heart failure requires the following

1. heart failure with reduced ejection fraction ( A 'reduced' ejection fraction (EF) defined as EF <40%): the presence of symptoms and/or signs of HF
2. heart failure with preserved ejection fraction ( A 'preserved' EF defined as EF≥ 40%) requires the all of the followings: a) the presence of symptoms and/or signs of HF b) elevated levels of natriuretic peptides (defined as B-type natriuretic peptide (BNP) >100pg/ml and/or N terminal B-type natriuretic peptide (NT-proBNP) >300pg/ml) c) any structural heart disease (left atrial volume index ≥ 34 mL/m2, left atrial dimension ≥ 50 mm, posterior or septal wall thickness ≥ 11mm)

Exclusion Criteria:

* any severe condition limiting life less than 3 months
* the patient is not ready to contact by telephone at the end of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospitalized patients with acute decompensated heart failure
Sampling Method: Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
The incidence rate (%) of composite endpoint including cardiovascular mortality or hospital readmission | 12 months
  Cardiovascular mortality: death due to heart failure aggravation, arrhythmia, cerebrovascular events, myocardial infarction.
  Hospital readmission: any readmission

SECONDARY OUTCOMES:
The incidence rate (%) of all cause mortality | 12 months
  Any death after enrollment
The incidence rate (%) of cardiovascular mortality | 12 months
  Death due to heart failure aggravation, arrhythmia, cerebrovascular events, myocardial infarction.
The incidence rate (%) of hospital readmission | 12 months
  Any readmission after discharge
The incidence rate (%) of hospital readmission due to heart failure aggravation | 12 months
  Readmission due to heart failure aggravation after discharge
The incidence rate (%) of cerebrovascular events | 12 months
  Stroke or intracranial hemorrhage
The incidence rate (%) of acute coronary syndrome | 12 months
  Unstable angina or myocardial infarction

CONTACTS AND LOCATIONS:
Overall Officials: Byung-Su Yoo, MD, PhD, Principal Investigator — Wonju College of Medicine, Yonsei University
Locations (1):
- Yonsei University Wonju College of Medicine, Wŏnju, Gangwondo, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ponikowski P, Voors AA, Anker SD, Bueno H, Cleland JG, Coats AJ, Falk V, Gonzalez-Juanatey JR, Harjola VP, Jankowska EA, Jessup M, Linde C, Nihoyannopoulos P, Parissis JT, Pieske B, Riley JP, Rosano GM, Ruilope LM, Ruschitzka F, Rutten FH, van der Meer P; Authors/Task Force Members; Document Reviewers. 2016 ESC Guidelines for the diagnosis and treatment of acute and chronic heart failure: The Task Force for the diagnosis and treatment of acute and chronic heart failure of the European Society of Cardiology (ESC). Developed with the special contribution of the Heart Failure Association (HFA) of the ESC. Eur J Heart Fail. 2016 Aug;18(8):891-975. doi: 10.1002/ejhf.592. Epub 2016 May 20. No abstract available. PMID 27207191
- [Background] Lee SE, Lee HY, Cho HJ, Choe WS, Kim H, Choi JO, Jeon ES, Kim MS, Kim JJ, Hwang KK, Chae SC, Baek SH, Kang SM, Choi DJ, Yoo BS, Kim KH, Park HY, Cho MC, Oh BH. Clinical Characteristics and Outcome of Acute Heart Failure in Korea: Results from the Korean Acute Heart Failure Registry (KorAHF). Korean Circ J. 2017 May;47(3):341-353. doi: 10.4070/kcj.2016.0419. Epub 2017 May 25. PMID 28567084
- [Background] Lee SE, Cho HJ, Lee HY, Yang HM, Choi JO, Jeon ES, Kim MS, Kim JJ, Hwang KK, Chae SC, Seo SM, Baek SH, Kang SM, Oh IY, Choi DJ, Yoo BS, Ahn Y, Park HY, Cho MC, Oh BH. A multicentre cohort study of acute heart failure syndromes in Korea: rationale, design, and interim observations of the Korean Acute Heart Failure (KorAHF) registry. Eur J Heart Fail. 2014 Jun;16(6):700-8. doi: 10.1002/ejhf.91. Epub 2014 May 2. PMID 24797348
- [Background] Kempf T, Eden M, Strelau J, Naguib M, Willenbockel C, Tongers J, Heineke J, Kotlarz D, Xu J, Molkentin JD, Niessen HW, Drexler H, Wollert KC. The transforming growth factor-beta superfamily member growth-differentiation factor-15 protects the heart from ischemia/reperfusion injury. Circ Res. 2006 Feb 17;98(3):351-60. doi: 10.1161/01.RES.0000202805.73038.48. Epub 2006 Jan 5. PMID 16397141
- [Background] Kempf T, Zarbock A, Widera C, Butz S, Stadtmann A, Rossaint J, Bolomini-Vittori M, Korf-Klingebiel M, Napp LC, Hansen B, Kanwischer A, Bavendiek U, Beutel G, Hapke M, Sauer MG, Laudanna C, Hogg N, Vestweber D, Wollert KC. GDF-15 is an inhibitor of leukocyte integrin activation required for survival after myocardial infarction in mice. Nat Med. 2011 May;17(5):581-8. doi: 10.1038/nm.2354. Epub 2011 Apr 24. PMID 21516086
- [Background] Xu XY, Nie Y, Wang FF, Bai Y, Lv ZZ, Zhang YY, Li ZJ, Gao W. Growth differentiation factor (GDF)-15 blocks norepinephrine-induced myocardial hypertrophy via a novel pathway involving inhibition of epidermal growth factor receptor transactivation. J Biol Chem. 2014 Apr 4;289(14):10084-94. doi: 10.1074/jbc.M113.516278. Epub 2014 Feb 19. PMID 24554716
- [Background] Dominguez-Rodriguez A, Abreu-Gonzalez P, Avanzas P. Relation of growth-differentiation factor 15 to left ventricular remodeling in ST-segment elevation myocardial infarction. Am J Cardiol. 2011 Oct 1;108(7):955-8. doi: 10.1016/j.amjcard.2011.05.028. Epub 2011 Jul 23. PMID 21784389
- [Background] Kempf T, von Haehling S, Peter T, Allhoff T, Cicoira M, Doehner W, Ponikowski P, Filippatos GS, Rozentryt P, Drexler H, Anker SD, Wollert KC. Prognostic utility of growth differentiation factor-15 in patients with chronic heart failure. J Am Coll Cardiol. 2007 Sep 11;50(11):1054-60. doi: 10.1016/j.jacc.2007.04.091. Epub 2007 Aug 24. PMID 17825714
- [Background] Cotter G, Voors AA, Prescott MF, Felker GM, Filippatos G, Greenberg BH, Pang PS, Ponikowski P, Milo O, Hua TA, Qian M, Severin TM, Teerlink JR, Metra M, Davison BA. Growth differentiation factor 15 (GDF-15) in patients admitted for acute heart failure: results from the RELAX-AHF study. Eur J Heart Fail. 2015 Nov;17(11):1133-43. doi: 10.1002/ejhf.331. Epub 2015 Sep 3. PMID 26333529
- [Background] Redfield MM. Heart Failure with Preserved Ejection Fraction. N Engl J Med. 2016 Nov 10;375(19):1868-1877. doi: 10.1056/NEJMcp1511175. No abstract available. PMID 27959663
- [Background] Chan MM, Santhanakrishnan R, Chong JP, Chen Z, Tai BC, Liew OW, Ng TP, Ling LH, Sim D, Leong KT, Yeo PS, Ong HY, Jaufeerally F, Wong RC, Chai P, Low AF, Richards AM, Lam CS. Growth differentiation factor 15 in heart failure with preserved vs. reduced ejection fraction. Eur J Heart Fail. 2016 Jan;18(1):81-8. doi: 10.1002/ejhf.431. Epub 2015 Oct 25. PMID 26497848
- [Derived] Cho DH, Son JW, Lee CJ, Choi J, Kim MN, Lee JH, Lee S, Yang DH, Cho HJ, Choi JO, Kim EJ, Choi DJ, Yoo BS. Prognostic Value of Short-Term Follow-up of Multiple Biomarkers After Discharge in Hospitalized Patients With Acute Heart Failure (POSTBIO-HF): Rationale and Study Design. Int J Heart Fail. 2022 Apr 4;4(2):110-116. doi: 10.36628/ijhf.2022.0005. eCollection 2022 Apr. PMID 36263107